CLINICAL TRIAL: NCT00859690
Title: Regulation of Vascular Thrombosis in Sleep Apnea
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 0901010175; Robert Wood Johnson Foundation
Record Dates: First submitted 2009-03-10; First posted 2009-03-11 (Estimated); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive Sleep Apnea; Thrombosis; Adenosine Deaminase; Sleep Disorder
MeSH Terms: conditions — Sleep Apnea, Obstructive; Thrombosis; Sleep Wake Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — A total of 15ml (approximately 1 tablespoon) of whole blood will be collected from each subject during his or her out-patient office visit. This sample will be retained for genomic analysis
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Sleep Disorder - Sleep Apnea: Subjects determined by a clinically indicated overnight sleep study (Nocturnal Polysomnography) to have Obstructive Sleep Apnea (OSA).
- Sleep Disorder - Not Sleep Apnea: Subjects determined by a clinically indicated overnight sleep study (Nocturnal Polysomnography) to have a sleep disorder other than Obstructive Sleep Apnea (OSA).

SUMMARY:
Sleep Apnea is a prevalent condition that has been increasingly diagnosed in the adult population and is now considered an independent risk factor for the development of cardiovascular disease. A better understanding of the mechanisms associated with the development of cardiovascular disease in sleep apnea is needed.

This research will investigate the function of the adenosine deaminase (ADA) in subjects with sleep disorders. This enzyme is responsible for metabolizing adenosine, a neuromodulator that is released during periods of sleep apnea and that has been found to promote vascular thrombosis. There are multiple types of ADA that are genetically determined and have different levels of function. Those different forms of this enzyme may determine groups that are more susceptible to the development of thrombosis. Given the known association between sleep apnea and thrombosis, this study will determine if polymorphisms of this enzyme are differentially found in subjects with sleep apnea as compared to other sleep disturbances. The overall objective of this experiment is to assess the presence of ADA polymorphisms in sleep apnea.

DETAILED DESCRIPTION:
Obstructive Sleep Apnea (OSA) is a prevalent condition that has been increasingly diagnosed in the adult population and is now considered an independent risk factor for the development of cardiovascular disease. More specifically, OSA has been linked with thrombosis, or the formation of clots in the blood vessels which can lead to heart attack or stroke. A better understanding of the mechanisms associated with thrombosis and the development of cardiovascular disease in patients with obstructive sleep apnea is needed.

This research will investigate the function of the enzyme adenosine deaminase (ADA) in subjects with sleep disorders. ADA is responsible for metabolizing adenosine, a neuromodulator that is released during periods of sleep apnea and that has been found to promote vascular thrombosis. There are multiple types of ADA that are genetically determined and have different levels of function. Those different forms of this enzyme may determine groups that are more susceptible to the development of thrombosis. Given the known association between sleep apnea and thrombosis, this study will determine if polymorphisms of this enzyme are differentially found in subjects with sleep apnea as compared to other sleep disturbances.

A total of 60 subjects presenting for the evaluation of sleep disorders to the Weill Cornell Pulmonary Associates and the Cornell Center for Sleep Medicine practices will be offered participation in this study. The subjects with sleep apnea will be ethnically matched to the subjects with sleep disorders other than sleep apnea (controls). Once written informed consent is obtained by the Principal Investigator, venipuncture will be performed in the office by a trained phlebotomist. A total of 15 ml (approximately 1 tablespoon) of blood will be collected. The patient will be monitored for ten minutes following the blood draw to ensure adequate hemostasis. The blood samples will be utilized for DNA sequencing and determination of adenosine deaminase genotype and phenotype.

Information from clinically indicated overnight sleep studies performed within 6 months of (prior or after) the visit will be used to categorize subjects into groups (sleep apnea vs. sleep disorder other than sleep apnea).

ELIGIBILITY:
Inclusion Criteria:

* 21 years or older
* Patient of the Weill Cornell Pulmonary Associates and Cornell Center for Sleep Medicine practices
* Clinically indicated for an overnight sleep study within six months prior to or after the outpatient office visit

Exclusion Criteria:

* Pregnancy

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from patients presenting for sleep disorders at the Weill Cornell Pulmonary Associates / Cornell Center for Sleep Medicine practices at New York-Presbyterian Hospital in New York City.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2009-03; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
ADA gene sequence | Determined after outpatient blood draw

CONTACTS AND LOCATIONS:
Overall Officials: Ana C Krieger, MD, MPH, Principal Investigator — Weill Medical College of Cornell University